CLINICAL TRIAL: NCT04612829
Title: Open-Label, Randomized, Active Controlled, Single Arm, Study to Ensure the Efficacy and Safety of Medistus Antivirus Lozenges in Mild to Moderate Acute Pharyngitis or Sore Throat or Strep Throat.
Brief Title: To Check Effectiveness of Medistus Antivirus Lozenges for Cough
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nutrin GmbH (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NUTRIN002
Record Dates: First submitted 2020-08-21; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Throat Infection; Pharyngitis; Sore Throat
Keywords: medistus; nutrin gmbh; throat infection; Pharyngitis; Antivirus
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention- Medistus Antivirus Lozenges (Experimental): A blend of Kistosyn Extract with Gum Arabic 1 Lozenge after every 2 hours, 5 times a day. Mode of Administration: Oral Duration of Treatment: 5 days
  Interventions: Device: Medistus Antivirus Lozenges

INTERVENTIONS:
Device: Medistus Antivirus Lozenges — A blend of Kistosyn Extract with Gum Arabic

SUMMARY:
A thraot infection sometimes called pharyngitis can be either a bacterial or a viral infection leading to inflammation of the tissues of the throat that causes redness, pain and swelling of the walls and structure of the throat.

The throat or Pharynx is the tube like structure that carries both food to the oesophagus and air to your wind pipe (called the larynx). Infective agents of the throat most often enters through the month or nose. Many of these infections are viral, other can be caused by bacteria such as Streptococcus Pyogenes, or Group A streptococcus.

Symtoms of throat infections most commonly includes pain and a sensation of heat in the throat or Pharynx.

Viral infections accounts for approx. 70% of all pharyngitis. Rhinovirus is the most common cause of viral infections. The other common causes of viral infections in descending order are corona virus, adeno virus, para influenza, and influenza virus. Viral infections are more common during the winter month with the exception of adeno viruses which occur year round.

Viral Pharyngitis is spread through similar mechanism as other viral infections. Hand to mouth contact, contact with oral secretions, and sharing common utensils, all contributes to viral spread.

Prevention of the spread of diseases is based on frequent hand washing, and clinical symptoms of different viruses are more prevalent during certain seasons. Coryza, conjectivitis, malease, or fatigue, hoarseness, and low grade fever such as the presence of viral phayngitis. Subjects with viral pharyngitis can also have atypical symptoms such as mouth breathing, nausea, abdominal pain, and diarrhoea.

Medistus Antivirus is a medical device product with a noble impact. Kistosyn 100 extract contains polyphenols, and with the help of gum arabic, it forms a protective film over the mouth and throat mucus membranes. This protective Barrier lead to a physical (mechanical) barrier against viruses and bacteria which prevent their penetration into body cells, and their further propagation. Due to this physical effect, resistance development is not possible.

ELIGIBILITY:
Inclusion Criteria:

* Patient with mild to moderate acute Pharyngitis or sore throat or strep throat
* Voluntarily signed informed consent for participation in this clinical study
* Compliance by the patient seems guaranteed, and the patient seems to be able to understand and complete the patient diary.

Exclusion Criteria:

* Severe respiratory tract infection (pneumonia, bronchitis or laryngitis)
* Oro-pharyngeal paresthesia or mycosis
* Severely traumatised and/or very severe oromucosal inflammation
* Tonsillopharyngectomy
* Peritonsillar abscess
* Long term use (≥ 3 times per week within the last month or regular intake within the last 3 months before randomisation) of antiinflammatory drugs- Any long-acting or slow release analgesic intake including NonSteroidal Anti-Inflammatory Drugs(NSAIDs)within 24 hours before randomisation (e.g. piroxicam or naproxen)
* Any anti-inflammatory drugs intake by systemic route within 12 hours before assigning
* Any paracetamol intake within 6 hours before randomisation
* Any cold medication (decongestant, antihistamine, expectorant, antitussive) within 6 hours before randomisation
* Any topical throat medication intake containing or not a local oral anaesthetic such as lozenge, spray, mouth rinse within 4 hours before recruitment
* Heavy smokers (>20 cigarettes/day)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2017-10-15 (Actual); Study Completion 2017-10-15 (Actual)

PRIMARY OUTCOMES:
To assess the cough episodes count | 5 days
  data collection on visit 2 from the subject for improvement in cough count
Throat pain assessment | 5 days
  on severity scale of 0-4
Redness of throat | 5 days
  on severity scale of 0-4
Swelling assessment | 5 days
  on severity scale of 0-4

CONTACTS AND LOCATIONS:
Overall Officials: Puneet Mittal, Study Director — Mittal Global Clinical Trial Services
Locations (1):
- Arogyam Superspeciality Hospital, Nagpur, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No
No plan to share